CLINICAL TRIAL: NCT01837875
Title: Intervention to Improve Quality of Life for African-AmericaN Lupus Patients (IQAN)
Brief Title: Intervention to Improve Quality of Life in African American Lupus Patients
Acronym: IQAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: IQAN; 1K01AR060026 (NIH)
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Depression; Systemic Lupus Erythematosus
Keywords: Intervention; Quality of life; African American; Stress
MeSH Terms: conditions — Depression; Lupus Erythematosus, Systemic | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Mailed informational literature
- Set Menu (Active Comparator): Intervention: Enrollment in a local Chronic Disease Self-Management program (CDSMP) and monthly follow up calls to gauge progress and comfort
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP)
- Intervention (Experimental): Intervention: Each individualized intervention plan (IIP) will include 1-4 options, including a mail-delivered arthritis kit, addition and access to a listserv, participation in a support group, and enrollment in local self-management program(s).
  Interventions: Behavioral: Chronic Disease Self-Management Program (CDSMP); Behavioral: Mail-delivered arthritis kit; Behavioral: Support group; Behavioral: Listserv

INTERVENTIONS:
Behavioral: Chronic Disease Self-Management Program (CDSMP) — The Chronic Disease Self-Management Program (CDSMP) is a 2.5 hour workshop given weekly for six weeks. People with different chronic health problems attend together and support one another in making positive changes in their health. Workshops are facilitated by two trained leaders, one or both of whom are non-health professionals with a chronic disease themselves. It is the process in which the program is taught that makes it effective. Classes are highly participative, and mutual support builds the participants' confidence in their ability to manage their health and maintain active and fulfilling lives.
  Arms: Intervention; Set Menu
Behavioral: Mail-delivered arthritis kit — The Arthritis Self-Management Tool Kit contains 1) a "Self Test" to help participants determine how arthritis affects their lives and self-tailor the use of the Tool Kit, including items related to pain, fatigue, physical limitations, and health worries; 2) information sheets: Working with Your Doctor and the Health Care System; Exercise; Medications; Healthy Eating; Fatigue and Pain Management; Finding Community Resources; and Dealing with One's Emotions; 3) information sheets on key process components of the ASMP: Action Planning, Problem Solving, Deciding What to Try, and Individualizing an Exercise Program; 4) The Arthritis Helpbook; 5) audio relaxation and exercise compact discs (CDs); and 6) an audio CD of all material printed on the information sheets.
  Arms: Intervention
Behavioral: Support group — Interested participants will be referred to the "Lupus: Listening and Learning Group", a Charleston-based support group affiliated with the Lupus Foundation of America (LFA). One to two LFA-trained facilitators implement the group. The meeting format generally includes a specific discussion topic or an informative presentation such as by a medical or counseling professional, pharmacist, or lupus researcher. This program is followed by time within the group for further interaction and support among the attendees who wish to participate. The Lupus: Listening and Learning Group is open to all lupus patients, family members, friends and supporters, and there is no pre-registration or fee involved.
  Arms: Intervention
Behavioral: Listserv — A project listserv will be established to link all intervention participants to facilitate exchange of coping strategies, pose questions, and share preferred educational resources or any other information relative to their everyday and disease-specific experiences and/or participation in the project. Participants will be provided with a URL, from which they will be able to subscribe to the listserv. Once subscribed, they will be able to post and receive messages, managed by a listserv moderator, who will be responsible for distribution to listserv members as appropriate. Participants will have the option to unsubscribe at any time.
  Arms: Intervention

SUMMARY:
The goal of the proposed project is to enhance the Principal Investigator's research ability to conduct behavioral interventions for people with lupus. This includes intervention design, implementation, data collection and data analysis. The Intervention to Improve Quality of life for African-AmericaN lupus patients (IQAN) Project is designed to examine whether a uniquely tailored intervention program can improve quality of life, decrease indicators of depression, and reduce perceived and biological indicators of stress in African American lupus patients. This study builds on three decades of work conducted in the field of arthritis self-management but differs in that the intervention mode, the disease (lupus), and the study population (African-Americans) are unstudied or understudied. The IQAN Project will use the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) model as its theoretical framework. This program has three specific aims. The first aim seeks to design a three armed randomized, wait list controlled trial that employs a patient-centered 'a-la-carte' approach that offers subjects a variety of modes of interaction, allowing them to choose as many or few as they wish. The second aim is to assess the intervention, using the RE-AIM model framework. The third aim, to be achieved before the first aim, is to use previously collected data to characterize patient-centric barriers to care in African-American lupus patients, in order to identify trends in patient needs and desires, as well as correlates of non-response and non-compliance that can be used in the development and refinement of the intervention.

DETAILED DESCRIPTION:
The intervention will be coordinated by an Intervention Coordinator, with assistance from local/MUSC Study Coordinators. A unique 'a-la-carte' self-management program will be offered to 50 African-American lupus patients participating in an ongoing SLE Clinic Database Project at MUSC. The Intervention Coordinator will work with each participant in the intervention arm to create an individualized intervention plan (IIP). Each IIP will include 1-4 options, including a mail-delivered arthritis kit, addition and access to a listserv, participation in a support group, and enrollment in local self-management program(s). Due to the nature of the IIP, the proposed intervention will inherently vary by participant. A 'set menu' control group of 50 lupus patients will be offered a standardized chronic disease self-management program only, and a control group of 50 lupus patients will receive usual care (UC), void of intervention components. Validated measures of stress, depression, and quality of life will be collected in all patients in each condition before and after intervention activities. To ensure intervention integrity, discrete components will follow written protocols and peer leaders will complete a standardized checklist for each session/encounter.

ELIGIBILITY:
Inclusion Criteria:

* formal diagnosis of lupus
* Black or African American

Exclusion Criteria:

* Younger than 18 years
* CNS/neuropsychiatric lupus and/or dementia
* participation in a chronic disease self management program in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Two years

SECONDARY OUTCOMES:
Disease Activity | Two years

OTHER OUTCOMES:
Stress | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Partnerships to Eliminate Health Disparities, University of South Carolina, Columbia, South Carolina, United States

REFERENCES:
- [Derived] Williams EM, Lorig K, Glover S, Kamen D, Back S, Merchant A, Zhang J, Oates JC. Intervention to Improve Quality of life for African-AmericaN lupus patients (IQAN): study protocol for a randomized controlled trial of a unique a la carte intervention approach to self-management of lupus in African Americans. BMC Health Serv Res. 2016 Aug 2;16(a):339. doi: 10.1186/s12913-016-1580-6. PMID 27485509